CLINICAL TRIAL: NCT04401137
Title: A Single Center, Randomized, Double Blind, Placebo Controlled, Dose Escalation Clinical Trial to Evaluate Pharmacokinetic/Pharmacodynamic Characteristics and Safety of QDX After Single Oral Administration in Healthy Korean Male Subjects
Brief Title: The Evaluation of Pharmacokinetic/Pharmacodynamic Characteristics and Safety of QDX in Healthy Korean Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: QDX001
Record Dates: First submitted 2020-05-14; First posted 2020-05-26 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-05

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Topiramate
- QDX 25 (Experimental)
  Interventions: Drug: Topiramate
- QDX 50 (Experimental)
  Interventions: Drug: Topiramate
- QDX 100 (Experimental)
  Interventions: Drug: Topiramate
- QDX 200 (Experimental)
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Topiramate — Topiramate

SUMMARY:
To evaluate pharmacokinetic/pharmacodynamic characteristics and safety of QDX after single oral administration in healthy Korean male subjects

ELIGIBILITY:
Inclusion Criteria:

* Participants who have fully understood this clinical trial via detailed explanation, are willing to voluntarily participate in this study, and agree to give written informed consent which is confirmed from IRB.
* Healthy male participants aged between 19 and 45 years at screening
* Those whose body weight is over 50kg, and BMI is between 18.0 and 27.0
* Participants who have demonstrated at least a 100 percent (%) increase in dermal blood flow in 30 minutes after capsaicin challenge as part of the screening procedures.

Exclusion Criteria:

* Those who have a clinically significant disease of liver, kidney, digestive, respiratory, endocrine, neurologic, blood/tumor, cardiovascular system, or history of those diseases
* Those who have a history of hypersensitivity or clinically significant hypersensitivity reactions to drugs (containing Topiramate etc.)
* Those who have a hereditary galactose intolerance, lapp lactase deficiency or glucose-galactose malabsorption syndrome
* Those who have irritating skin, wounds, eczema, and wounds on the area where capsaicin is applied

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
The Capsaicin-Induced Dermal Blood Flow (DBF) | Pre-dose(-2 hour), 2 hour, 4 hour, 8 hour, 24 hour post-dosing on Day1
  Change from Baseline in Dermal Blood Flow Induced by QDX Compared to Placebo
Area Under the Plasma Concentration-time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUC[0-T]) | Pre-dose(-2 hour), 2 hour, 4 hour, 8 hour, 12hour, 24 hour post-dosing on Day1
  Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration.
Area Under the Plasma Concentration-time Curve From Time Zero to the Time of Last Quantifiable Plasma Concentration (AUClast) | Pre-dose(-2 hour), 2 hour, 4 hour, 8 hour, 12hour, 24 hour post-dosing on Day1
  Area under the plasma concentration-time curve from time zero to the last quantifiable concentration.
Maximum Observed Plasma Concentration (Cmax) | Pre-dose(-2 hour), 2 hour, 4 hour, 8 hour, 12hour, 24 hour post-dosing on Day1
  Maximum observed plasma concentration following drug administration from the raw plasma concentration-time data.
Time to Reach Maximum Plasma Concentration (Tmax) | Pre-dose(-2 hour), 2 hour, 4 hour, 8 hour, 12hour, 24 hour post-dosing on Day1
  Tmax was defined as the time required to reach maximum observed plasma concentration.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Dept. of Clinical Pharmacology, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided